CLINICAL TRIAL: NCT00065676
Title: Inhibition of Intestinal Glucose Absorption by the Bioflavonoid Quercetin in the Obese and in Obese Type 2 Diabetics
Brief Title: Investigating the Use of Quercetin on Glucose Absorption in Obesity, and Obesity With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 030256; 03-DK-0256
Record Dates: First submitted 2003-07-30; First posted 2003-07-31 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-01-22

CONDITIONS: Obesity; Diabetes
Keywords: Hyperglycemia; Hyperinsulinemia; OGTT; GLUT2; Post-Prandial; Type 2 Diabetes; Obesity
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Hyperglycemia; Hyperinsulinism; Diabetes Mellitus, Type 2 | interventions — Quercetin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 gram quercetin (Experimental): 1 gram quercetin with 6 hour OGTT
  Interventions: Other: Quercetin
- 2 grams quercetin (Experimental): 2 gram quercetin with 6 hour OGTT
  Interventions: Other: Quercetin
- placebo (Experimental): placebo with 6 hour OGTT
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Quercetin — 1 or 2 grams of quercetin or placebo will be given while patients undergo 6-hour OGTT
  Arms: 1 gram quercetin; 2 grams quercetin
Other: Placebo
  Arms: placebo

SUMMARY:
Quercetin is a compound naturally found in various foods. It may have some role in the treatment of obesity and diabetes.

The purpose of this study is to investigate research volunteers with obesity or obesity with type 2 diabetes to determine whether quercetin affects the way glucose is absorbed by the body.

Thirty two participants aged 19 to 65 who are considered to be medically obese or obese with type 2 diabetes will be enrolled in this study. Before the onset of treatment, they will undergo a medical history, physical exam, blood work, and urinalysis. During the study, participants will be given an oral glucose tolerance test three times; during these tests they will receive 1 or 2 grams of quercetin, or placebo. Researchers will collect blood samples and analyze the effect of the treatment on blood glucose.

DETAILED DESCRIPTION:
Postprandial hyperglycemia and the resultant hyperinsulinemia contribute to the cardiovascular complications seen in obesity and in type 2 diabetes. Epidemiological studies suggest that slow absorption of carbohydrates dampens glucose and insulin peaks, and reduces cardiovascular morbidity. The polyphenol quercetin is the most abundant flavanoid in plant-derived foods, and is sold as a dietary supplement. In vitro, quercetin is a potent and reversible inhibitor of glucose transport by the intestinal glucose transporter GLUT2. In vivo quercetin inhibits post absorptive glucose peaks in obese, diabetic rats. We hypothesize that quercetin blunts intestinal glucose absorption in humans, and attenuates postprandial hyperglycemia. We propose to test, in a double blind placebo controlled study, whether coadministration of 1 or 2 grams of quercetin with glucose will reduce plasma glucose concentrations during a 6 hour oral glucose tolerance test with 3 to 6 grams of 3-O-methyl glucose (3OMG) in non-diabetic obese subjects and in obese type 2 diabetic subjects. The glucose dose may be varied from 0 to 100 grams to better understand the competition between 3OMG and glucose. 3OMG is a non-metabolizable glucose analogue and is excreted unaltered in urine. 3OMG is not found in food and thus glucose absorption can be studies easily without the problem of a high baseline value. The use of 3OMG will provide a more accurate and true measures of glucose absorption. Study subjects will be 19 - 65 years with a body mass index greater than or equal to 30, without complications of diabetes, or on any medication other than oral hypoglycemic agents and aspirin. We will study 16 obese non diabetic subjects and 16 obese type 2 diabetics. Each subject will have 3 oral glucose tolerance tests, and will serve as his or her own control. We will compare the peak plasma glucose concentrations achieved during oral glucose tolerance tests and the area under the curve of plasma glucose to determine whether quercetin inhibits glucose absorption in humans. Such inhibition may partially explain the protective effects of plant derived foods on cardiovascular disease, and enable us to use quercetin or related compounds to dampen intestinal glucose absorption. We will also measure quercetin concentrations in the plasma, in circulating white blood cells and in urine to determine quercetin pharmacokinetics. Additionally, to determine the optimal 3OMG dose, we will study the absorption of glucose and 3OMG, without quercetin, in 12 non-diabetic obese subjects and 12 lean subjects to serve as controls.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects to be recruited for the study will be male and female subjects between the ages of 18 and 65, able to give informed consent, with mild to moderate type 2 diabetes (such that fasting blood sugar <200mg/dl or HbA1C < 8.5), in otherwise good general health, with no other significant illnesses, blood pressure <=160/90 mmHg with or without medication, with no known severe target organ damage. End organ damage includes the following: proliferative retinopathy, serum creatinine >2, ischemic heart disease, congestive heart failure, known gastroparesis, peripheral vascular disease and severe peripheral neuropathy. Diabetic subjects must have a BMI greater than or equal to 30. Subjects will be taken off hypoglycemic agents for 3 to 7 days prior to each part of the study. This is to remove a confounding factor that may affect blood glucose concentrations attained during the OGTT, independent of the effect of quercetin. Whether these oral hypoglycemic agents have physiologically significant interaction with quercetin is not known. Severity of diabetes and biological duration of action of the drug will determine when to initiate this hold (from 3 to 7 days prior to OGTT). During the time that the subjects are off oral hypoglycemic agents, they will monitor their fasting blood glucose daily by glucometer. Therefore, for subjects with diabetes, only those subjects who self-monitor blood glucose are eligible for inclusion. If the fasting blood glucose in the morning exceeds 300 mg/dl, the subject will be withdrawn from the study and appropriate therapy resumed. Obese volunteers, with a BMI greater than or equal to 30, must be in good health, with no known illness. Healthy, normal weight subjects (BMI <25) will also be recruited as control subjects for the sampling study without querecetin. An upper age limit of 65 years was chosen to minimize renal toxicity of quercetin, as GFR declines with age and quercetin might produce mild though reversible renal impairment.

EXCLUSION CRITERIA:

Exclusion criteria will include the following: significant digestive abnormalities such as malabsorption or chronic diarrhea; significant organ malfunction including (but not limited to) liver disease, pulmonary disease, ischemic heart disease, heart failure, stroke, peripheral vascular disease, hypertension (BP >160/90), and anemia (hematocrit < 30); other serious or chronic illness; history of serious or chronic illness; any significant complications from diabetes such as kidney damage (renal insufficiency, serum creatinine >2), eye damage (proliferative retinopathy), severe diabetic neuropathy, coronary artery disease, or symptomatic peripheral vascular disease; smoking; alcohol or drug abuse; smokers; pregnancy (a urine pregnancy test will be performed on all women with reproductive age before each part of the study); lactation; positive HIV or hepatitis (B or C) screening tests (subjects will be notified of these test results). Diabetic subjects who choose not to self-monitor glucose daily by glucometer will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-04-30 (Actual); Primary Completion 2015-12-21 (Actual); Study Completion 2021-08-06 (Actual)

PRIMARY OUTCOMES:
Does quercetin effect glucose absorption | End of study
  Reduction in plasma glucose concentrations during 6-hour oral glucose tolerance test with 1 gram quercetin vs 2 grams quercetin vs placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Levine, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Mooradian AD, Thurman JE. Drug therapy of postprandial hyperglycaemia. Drugs. 1999 Jan;57(1):19-29. doi: 10.2165/00003495-199957010-00003. PMID 9951949
- [Background] Gavin JR 3rd. Pathophysiologic mechanisms of postprandial hyperglycemia. Am J Cardiol. 2001 Sep 20;88(6A):4H-8H. doi: 10.1016/s0002-9149(01)01830-6. PMID 11576519
- [Background] Yanovski SZ, Yanovski JA. Obesity. N Engl J Med. 2002 Feb 21;346(8):591-602. doi: 10.1056/NEJMra012586. No abstract available. PMID 11856799
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2003-DK-0256.html